CLINICAL TRIAL: NCT00006468
Title: Phase III Study of An Optimized LV-5FU-Oxaliplatin Regimen in Metastatic Colorectal Cancer. C99-1.
Brief Title: Comparing Two Combination Chemotherapy Regimens in Treating Patients With Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068282; FRE-GERCOR-OPTIMOX-2000; EU-20034
Record Dates: First submitted 2000-11-06; First posted 2003-01-27 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2000-12

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; Fluorouracil; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: FOLFOX regimen
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which regimen of combination chemotherapy is more effective for metastatic colorectal cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two combination chemotherapy regimens in treating patients who have metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of intermittent high-dose oxaliplatin in combination with a simplified bimonthly regimen of leucovorin calcium (LV) and fluorouracil (5-FU) vs standard dose oxaliplatin in combination with the standard bimonthly regimen of LV and 5-FU in patients with metastatic colorectal cancer.
* Determine the time to treatment failure, tolerance, response rate, and overall survival in patients treated with these 2 regimens.
* Compare quality of life of these patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to treatment center, performance status (0-1 vs 2), and number of metastatic sites (1 vs more than 1). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive oxaliplatin IV over 2 hours on day 1, and leucovorin calcium IV over 2 hours followed by fluorouracil (5-FU) IV over 22 hours on days 1 and 2.
* Arm II: Patients receive oxaliplatin IV and leucovorin calcium IV over 2 hours followed by 5-FU IV over 46 hours beginning on day 1 for courses 1-6 and 19-24. For courses 7-18, patients receive leucovorin calcium IV followed by 5-FU IV as above beginning on day 1.

Courses repeat every 14 days in both arms in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, after courses 4 and 6, and every 6 courses thereafter.

Patients are followed monthly for 3 months and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 460 patients (230 per treatment arm) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed unresectable metastatic adenocarcinoma of the colon or rectum
* Bidimensionally measurable or evaluable disease outside previously irradiated area

  * No bone metastasis as target lesion
  * At least 1 cm if spiral CT scan OR
  * At least 2 cm if conventional CT scan
* No CNS metastasis
* No symptomatic ascites or pleural effusion that is not evacuated
* No total or partial bowel obstruction

PATIENT CHARACTERISTICS:

Age:

* 18 to 80

Performance status:

* ECOG 0-2
* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Alkaline phosphatase less than 5 times upper limit of normal (ULN)

Renal:

* Creatinine less than 3 times ULN
* No uncontrolled hypercalcemia

Cardiovascular:

* No uncontrolled congestive heart failure, angina pectoris, hypertension, or arrhythmias

Other:

* No peripheral sensory neuropathy
* No prior significant neurologic or psychiatric disorders
* No other malignancy within past 5 years except adequately treated carcinoma in situ of the cervix or basal or squamous cell skin carcinoma
* No active infection
* No other concurrent serious disease
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy for metastatic disease

Chemotherapy:

* Prior adjuvant chemotherapy allowed, provided progression-free interval of more than 6 months since end of last course
* No prior oxaliplatin or irinotecan
* No prior chemotherapy for metastatic disease
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No concurrent radiotherapy

Surgery:

* Concurrent surgery allowed

Other:

* At least 30 days since other prior investigational drugs
* No other concurrent investigational treatment
* No other concurrent antitumoral treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01

CONTACTS AND LOCATIONS:
Overall Officials: Aimery de Gramont, MD, Study Chair — Hopital Saint Antoine
Locations (1):
- Hopital Saint Antoine, Paris, France